CLINICAL TRIAL: NCT04750291
Title: Management of Popeye Sign With Botulinum Toxin After Tenotomy of the Long Head of the Biceps Tendon: a Double-blinded Randomized Controlled Trial
Brief Title: Management of Popeye Sign With Botulinum Toxin After Bicepstenotomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: AZ Delta (Other)
Responsible Party: Principal Investigator, Bert VanMierlo, Principal Investigator, AZ Delta
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12217
Record Dates: First submitted 2021-02-08; First posted 2021-02-11 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Popeye Syndrome
Keywords: tenotomy; long head of the biceps tendon; botulinum toxin
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Botulinum toxin (Experimental): Infiltration with botulinum toxin
  Interventions: Drug: Botulinum toxin type A
- Placebo (Placebo Comparator): Infiltration with placebo or sterile saline
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Botulinum toxin type A — 1 infiltration in the biceps muscle with botulinum toxin (100 IU)
  Arms: Botulinum toxin
Other: Placebo — 1 infiltration in the biceps muscle with placebo or sterile saline
  Arms: Placebo

SUMMARY:
Double-blinded randomized controlled trial with 20 people of whom 10 will receive a placebo infiltration and 10 an infiltration with botulinum toxin type A for cramping pain after arthroscopic tenotomy of the long head of the biceps tendon.

DETAILED DESCRIPTION:
Title: Management of Popeye sign with botulinum toxin after tenotomy of the long head of the biceps tendon: a double-blinded randomized controlled trial Précis: Double-blinded randomized controlled trial with 20 people. Randomization in 2 arms of 10 people. 3 visits will be planned with a meantime of 3 months after the infiltration with botulinum toxin type A (BTX-A) or placebo that will be administered at the 2nd visit.

Objective: The primary objective is to assess the effectiveness of an infiltration with botulinum toxin in the biceps muscle after tenotomy of the long head of the biceps tendon for pain and disability reduction.

Endpoint: The primary endpoint is a pain reduction as measured by the Visual Analogue pain scale (VAS) and a reduced disability as measured by the quick DASH (Disabilities of the Arm, Shoulder and Hand).

Population: 20 people who underwent an arthroscopic tenotomy of the long head of the biceps tendon and are having post-operative pain in the biceps muscle.

Phase: 4

Number of Sites enrolling participants: single center study in AZ Delta Roeselare

Description of Study Agent: botulinum toxin type A (Botox®) 100 International Units by intramuscular injection

Study Duration: From March 2021 till December 2022

Participant Duration: 3 months

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Have had arthroscopic tenotomy of the long head of the biceps tendon without rotator cuff repair, acromioclavicular joint resection or glenoid labrum repair
* Having bicipital pain that started after the tenotomy

Exclusion Criteria:

* under 18 years of age
* over 65 years of age
* pregnancy or lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-08-09 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Pain change | 3 months
  VAS score: Visual Analogue Scale score of 0 to 10 with 0 indicating no pain and 10 the worst pain imaginable
Disability change | 3 months
  quick DASH: Disabilities of the Arm, Shoulder and Hand 0 (no disability) to 100 (most severe disability)

CONTACTS AND LOCATIONS:
Overall Officials: Bert Vanmierlo, MD, Principal Investigator — Orthopedie Roeselare AZ Delta
Locations (1):
- AZ Delta, Roeselare, Belgium

IPD SHARING:
Plan to Share IPD: No